CLINICAL TRIAL: NCT03242590
Title: Validation of Dosing Regimen of Oral Testosterone Undecanoate (TU, LPCN 1021) in Hypogonadal Men.
Brief Title: Dosing Validation Study of Oral Testosterone Undecanoate (TU, LPCN 1021).
Acronym: DV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lipocine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPCN 1021-16-002
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral testosterone undecanoate, LPCN 1021 (Experimental): Oral testosterone undecanoate, LPCN 1021 225 mg TU two times a day.
  Interventions: Drug: LPCN 1021

INTERVENTIONS:
Drug: LPCN 1021 — Oral testosterone undecanoate

SUMMARY:
Multicenter, open-label, one treatment study evaluating the efficacy of LPCN 1021 in adult hypogonadal male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Serum total T below 300 ng/dL based on 2 consecutive blood samples obtained between 6 and 10 AM, on two separate days at approximately the same time of day, following an appropriate washout of current androgen replacement therapy.
2. Subjects should be diagnosed to be primary (congenital or acquired) or secondary hypogonadal (congenital or acquired).
3. Naïve to androgen replacement or has discontinued current treatment and completed adequate washout of prior androgen therapy. Washout must be completed prior to collection of baseline serum T samples to determine study eligibility.

Exclusion Criteria:

1. History of significant sensitivity or allergy to androgens, or product excipients.
2. Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up.
3. Abnormal prostate digital rectal examination (DRE) with palpable nodule(s).
4. Subjects with symptoms of moderate to severe benign prostatic hyperplasia.
5. Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis
6. Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus antibodies (HIV Ab).
7. History of gastric surgery, cholecystectomy, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
8. History of any clinically significant illness, infection, or surgical procedure within 1 month prior to study drug administration.
9. History of stroke or myocardial infarction within the past 5 years.
10. History of or current or suspected prostate or breast cancer.
11. History of untreated and severe obstructive sleep apnea.
12. History of long QT syndrome (QTc > 450) or unexplained sudden death in a first degree relative (parent, sibling, or child).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DelConte, MD, Study Director — Lipocine Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DelConte A, Papangkorn K, Kim K, Bruno BJ, Chidambaram N, Khera M, Goldstein I, Kohler TS, Miner M, Dobs AS, Patel MV. A new oral testosterone (TLANDO) treatment regimen without dose titration requirement for male hypogonadism. Andrology. 2022 May;10(4):669-676. doi: 10.1111/andr.13153. Epub 2022 Jan 18. PMID 34994093

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Testosterone Undecanoate, LPCN 1021
Started | 95
Completed | 95
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oral Testosterone Undecanoate, LPCN 1021
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 77
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 95
Baseline Testosterone Value (ng/dL) [Mean (Standard Deviation); unit: ng/dL] | 202 (74.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent of LPCN 1021-treated Subjects Who Achieve a Total Testosterone Average Concentration [Cavg] in the Normal Range
Description: The primary efficacy endpoint and analysis for this study was the percentage of LPCN 1021 treated subjects who had achieved a 24-hour average serum T concentration within the normal range of 300 to 1080 ng/dL at Visit 4, (Day 24 ± 4 days).
Time Frame: Following 24 days of treatment
Population: Safety Set
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Oral Testosterone Undecanoate, LPCN 1021
Number analyzed (Participants) | 95
Percent of participants | 80 [72 to 88]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Oral Testosterone Undecanoate, LPCN 1021
All-Cause Mortality (participants affected / at risk) | 0/95
Serious Adverse Events (participants affected / at risk) | 1/95
Other Adverse Events (participants affected / at risk) | 6/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Testosterone Undecanoate, LPCN 1021 (N=95)
Gastric Ulcer Hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Testosterone Undecanoate, LPCN 1021 (N=95)
Blood prolactin increased (Endocrine disorders) | 4 (4)
Blood FSH decreased (Endocrine disorders) | 1 (1)
Blood LH decreased (Endocrine disorders) | 1 (1)
PSA increased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT03242590/Prot_SAP_000.pdf